CLINICAL TRIAL: NCT07134647
Title: Effects of Video Animation-Assisted Inhaler Medication Education on Medication Adherence, Attack Frequency, and Dyspnea for Asthma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, SEDA ILGUN, PhD Student, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GAZİANTEP UN; Seda İlgün (Registry Identifier: Gaziantep University Health Sciences Institute Internal Medicine Nursing)
Record Dates: First submitted 2025-07-15; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Asthma Control Level

STUDY DESIGN:
Intervention Model Description: Before the training, the researcher will administer data collection forms to both groups using a face-to-face interview. The researcher will then provide a face-to-face "Video Animation-Assisted Inhaler Medication Education" to the patients in the intervention group. After the initial interview, all training sessions will be provided online via the training link, and patients will be contacted weekly to request a repeat session. Patients will receive weekly online reminders of the training sessions. Patients in the control group will not receive any interventions other than the clinic's routine procedures. Data collection tools will be administered simultaneously with the intervention group. The control group will receive video-assisted inhaler medication education at the end of the study, if they wish. The questionnaire and scales will be administered at the beginning of the study, on day 15, and at the end of week 4.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group will not receive training. The evaluation form will be administered simultaneously with the intervention group. At the end of the study, the patient will be shown the video once if they wish.
- INTERVENTION GROUP (Experimental): Patients in the intervention group will watch an educational video at the beginning of the study, on the 15th day, and at the 4th week.
  Interventions: Behavioral: video animation-supported inhaler medication training

INTERVENTIONS:
Behavioral: video animation-supported inhaler medication training — The training is presented not verbally but with the prepared "Video Animation Support"
  Arms: INTERVENTION GROUP

SUMMARY:
Asthma is a chronic airway inflammation characterized by recurrent attacks, airway hyperresponsiveness, mucus hypersecretion, and airway obstruction. It ranks 16th among the most serious diseases in terms of duration and severity of disability. The disease poses a significant social and economic burden and morbidity for families and the healthcare system. It is estimated that approximately 300 million people worldwide are affected by asthma, and this number is expected to reach 400 million by 2025. Symptoms, airflow limitation, and its degree vary significantly over time in asthma. These changes are generally influenced by various stimuli, such as the presence of allergies or irritants, physical activity, air changes, or respiratory infections. Therefore, proper management of asthma, which poses a significant problem for both patients and society, is crucial. The goals of asthma treatment are to provide symptom control, reduce exacerbations, and alleviate fixed airway obstruction and medication side effects. Oral, parenteral, and inhaled agents are currently used in treatment. Inhaled treatments offer advantages over other treatment methods because they deliver medications directly to the airways and accumulate there, resulting in a faster onset of action and fewer side effects due to the use of smaller doses. Because inhaled medication must reach the targeted airways for it to be effective, proper inhalation technique is as important as adherence to treatment. However, it is known that 70-80% of patients fail to use their inhalers correctly. Failure to use inhalers properly and correctly leads to ineffective treatment, uncontrolled disease, frequent attacks, increased medication use, hospitalizations, and increased costs. Therefore, the most fundamental element of asthma treatment is inhaler use training. In addition to providing information about the disease, the patient should be thoroughly and practically instructed on how and when to use asthma medications. However, studies conducted in our country have shown that the rate of inhaler use using the correct technique is quite low. However, asthma management education has been proven effective in improving asthma control and quality of life. Numerous studies confirm that the use of smartphone-based apps is a promising educational tool. Effective use of new mobile apps and smart technologies is also noted to be important in improving treatment adherence rates, improving inhaler technique, and improving asthma control. Therefore, this study aimed to evaluate the effects of video-animated inhaler medication education on medication adherence, seizure frequency, and dyspnea in asthmatic patients.

DETAILED DESCRIPTION:
Asthma is a disease characterized by recurrent airway obstruction that can impair patients' quality of life and mental well-being. Asthma, which has a high prevalence among chronic diseases, is a significant public health problem among respiratory diseases. It can occasionally cause increases in symptom frequency and severity and can be life-threatening. Disease control in asthma is defined as the degree to which various symptoms of asthma are reduced or eliminated with treatment. Uncontrolled asthma imposes a significant social and economic burden on asthma patients. The cornerstones of treatment are guideline-based medication regimens and asthma education programs aimed at equipping patients for effective self-management. Poor disease control in asthma can result from patients being prescribed inappropriate medications or using prescribed medications incorrectly. Airway obstruction, associated with narrowing of the airway lumen, the most characteristic feature of asthma, is reversible with bronchodilator therapy . For inhalation therapy, the patient's choice of device that is easy and accurate to use and the correct inhaler technique are crucial. Device selection not only increases the success of medication administration but also improves patient compliance and asthma control. Improper inhaler technique can lead to patients receiving inadequate medication doses. This not only limits medication effectiveness but can also lead to side effects. Furthermore, even if the patient uses the medication as prescribed, incorrect inhaler technique can lead to poor disease control. Education is crucial in preventing or managing these problems. Nurse educators, as part of their role as educators, can identify the patient's learning potential and, through training, ensure that the patient uses inhaled medications correctly, thus increasing treatment success. Studies have shown that inhaler device training has significant positive effects on the correct use of the device. Gregoriano C. et al. concluded in their study that correct medication inhalation has a positive impact on health status and lung function. A study by Al-Kharouf MS and colleagues concluded that video-based training is effective in improving inhaler technique over time, as well as improving disease control, medication adherence, and quality of life. However, it is known that 70-80% of patients fail to use their inhalers correctly. One study found that the incidence of nonadherence was 47.6% based on patient reports and 48.5% based on pharmacy records. Paske et al. concluded that approximately 70% of asthma patients use inhaled medications incorrectly, leading to decreased disease control, increased healthcare utilization, and increased costs. A study by Mortan et al. found that patients generally have poor inhaler technique, resulting in suboptimal asthma control. A meta-analysis found that the reduction in the likelihood of exacerbations was greatest in patients with 80% or greater adherence to treatment, but a reduction was also observed among those with greater than 50% adherence. These results suggest that greater emphasis should be placed on the educational component of treatment. The standard mode of inhaler technique training in many studies has been written materials or verbal instructions. Single-session verbal training has a temporary effect on improving inhaler technique. One-on-one training sessions that include physical demonstrations of inhaler use are significantly more effective than written training. However, several studies have clearly demonstrated that inhaler technique deteriorates if training is not repeated within 1 to 3 months of physical demonstration. It is emphasized that at least three training sessions are necessary to develop effective inhalation technique. Although technique improves after verbal training, this can lead to inadequacies over time and requires reinforcement with different educational strategies. Video training tools have been used since the early 2000s and are considered useful interventions for promoting medication adherence and behavioral changes in patients. These tools can account for different learning preferences by providing patients with visual and auditory information about their medications and can be used to reinforce the importance of medication adherence and high-risk medications.Video education tools can also be used to address common patient concerns and can be adapted to meet individual patient needs, including language and literacy levels. Therefore, the development of patient education videos is thought to be beneficial in improving patient outcomes. Based on these results, we planned to evaluate the effects of video animation-assisted inhaler medication education on medication adherence, seizure frequency, and dyspnea in asthmatic patients.

ELIGIBILITY:
Inclusion Criteria:

Patients who are:

* 18 years of age or older,
* Diagnosed with asthma for at least 6 months,
* Using at least one inhaler,
* No communication problems that would prevent them from participating in the study or receiving training,
* Literate,
* Have internet access at home or on their phone,
* Own and use a computer, tablet, or smartphone,
* Voluntarily agree to participate in the study

Exclusion Criteria:

Individuals who:

* Do not meet the inclusion criteria,
* Are unwilling to participate in the study,
* Do not own a computer, tablet, or smartphone,
* Have a psychiatric illness

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Video animation-assisted inhaler drug education has effects on drug compliance, attack frequency and dyspnea. | Each patient will be followed up for 30 days.
  Data were collected using a questionnaire, the mMRC Shortness of Breath Scale, the Asthma Control Test (ACT), and the Inhaler Compliance Scale. The mMRC Shortness of Breath Scale is a 5-point scale (0-4). A higher score indicates greater severity of dyspnea. The Asthma Control Test (ACT) is a 25-point scale. A higher score is considered good control. The Inhaler Compliance Scale is a 30-point scale. A higher score indicates good inhaler compliance. The mMRC Shortness of Breath Scale, the Asthma Control Test (ACT), and the Inhaler Compliance Scale were administered to both groups at the beginning of the study and at the end of the fourth week. After 3 sessions of training, the decrease in the mMRC Shortness of Breath Scale mean score and the increase in the Asthma Control Test (ACT) and Inhaler Compliance Scale mean score indicate that the training was effective. Student t, chi-square, Mann Whitney U and Kruskal Wallis tests were used to evaluate the data.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep Üniversitesi, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No